CLINICAL TRIAL: NCT06005272
Title: Mothers Working to Prevent Early Stillbirth Study 20-28
Acronym: MiNESS20-28
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: University of Birmingham (Other); University of Leicester (Other); University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Professor of Obstetrics, University of Manchester
Other Study IDs: 314658
Record Dates: First submitted 2023-05-09; First posted 2023-08-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Stillbirth and Fetal Death; Perinatal Death
MeSH Terms: conditions — Stillbirth; Fetal Death; Perinatal Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Recently pregnant women/people who have experienced baby loss during pregnancy, labour or shortly after birth between 20-28 weeks of pregnancy
  Interventions: Other: Questionnaire
- Controls: Individuals still pregnant at same gestational age
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Interviewer assisted completion of questionnaire.

SUMMARY:
This project aims to identify factors linked to pregnancy losses occurring between 20 and 28 weeks of pregnancy that can be modified by changing mother's behaviour or healthcare provision.

The death of a child before birth (also called stillbirth or miscarriage) has enduring psychological, social and economic effects for women, their families and wider society. In 2015, the stillbirth rate in the UK was higher than comparable countries. The UK government has committed to reduce stillbirths by 50% by 2025. Presently, stillbirths after 28 weeks of pregnancy have reduced by 16% but there has been no change in losses between 20 and 28 weeks of pregnancy with 1,600 losses estimated to occur at this stage of pregnancy each year.

Identification of modifiable causes of stillbirth was identified as a research priority by the Stillbirth Priority Setting Partnership which involved over 1,000 participants, one third of whom were bereaved parents. The investigators previously completed a study of 291 women who had a late stillbirth (after 28 weeks of pregnancy) and 733 women who had a live baby in 41 maternity units in the UK. This study identified factors linked to stillbirth which can be changed including the position women go to sleep in, cigarette smoking and caffeine consumption. In addition, the investigators previously found changes in mother's perception of baby's movements, whether women had tests for diabetes or whether women were exposed to domestic violence or stressful situations. These factors can be addressed by different care in pregnancy. Information from this study has been included in national and international guidelines that aim to reduce stillbirth.

The investigators will use the same study type to identify factors associated with pregnancy loss between 20 and 28 weeks of pregnancy (early stillbirth). The investigators have asked parents who have experienced the death of a baby at these stages of pregnancy about the design of the study, the questions that would be asked and how best to approach bereaved parents. This led us to include miscarriages from 20-22 weeks of pregnancy that are not usually "counted" in UK stillbirth statistics. The investigators will need 316 women with stillbirth between 20 and 28 weeks of pregnancy and 632 women with an ongoing live pregnancy to participate in the study. All women will complete a questionnaire about themselves, their diet, behaviours and sleep, their baby's movements and pregnancy care. The investigators will compare information between women who have early stillbirth and those who have a live birth to identify factors associated with stillbirth at less than 28 weeks of pregnancy. The study findings will be disseminated in collaboration with patient organisations using effective ways to reach pregnant women. The investigators anticipate the findings from this study will be included in clinical practice guidelines and rapidly translated into antenatal care.

DETAILED DESCRIPTION:
Research question What are the modifiable risk factors for early stillbirth (between 20-28 weeks' gestation)?

Background The NHS Long Term Plan sets a goal to reduce stillbirth by 50% by 2025 (from 2013 rates). Some progress has been made with reduction of stillbirths in late pregnancy (≥28 weeks' gestation). However, rates of early stillbirth (<28 weeks' gestation) remain intractable and new initiatives to reduce early stillbirth rates are needed to achieve this goal. Our previous study (MiNESS) informed about modifiable risk factors for stillbirth ≥28 weeks' gestation and were incorporated into national guidance to reduce stillbirth. However, there is an evidence gap related to modifiable risk factors for early stillbirth.

Aims and Objectives The overall aim of the study is to

1. Identify modifiable risk factors for early stillbirth that are amenable to public health campaigns or adaptation of antenatal care.

   The study will specifically,
2. Confirm or refute whether modifiable behavioural factors associated with late stillbirth are also independently associated with early stillbirth.
3. Explore interactions between maternal characteristics (especially those relating to health inequalities including ethnicity and socioeconomic deprivation), fetal factors (including fetal growth restriction, reduced fetal movements) and early stillbirth risk.
4. Determine differences in risk factor profiles by cause of death.

Methods This study uses a case-control design based upon that successfully used in the MiNESS study. The eligible population are women with a non-anomalous singleton pregnancy. "Cases" are women who have a stillbirth between 20+0 and 27+6 weeks' gestation and "Controls" are women who have an ongoing viable pregnancy at an equivalent gestational age. Controls will be randomly selected from participating maternity units' booking list at the appropriate week of pregnancy to match the unit's historic distribution of early stillbirths in a 1:2 (case:control) ratio. The study will recruit 316 cases and 632 controls; this gives 80% power to detect associations with an odds ratio ≥1.5. Participants will complete a researcher-administered questionnaire and relevant data will be extracted from medical records. Cases will be approached before hospital discharge, aiming to complete the research interview where possible within 3 weeks.

Unadjusted associations between early stillbirth and each exposure will be calculated. Logistic regression models, adjusted for confounding variables, will consider multiple exposures in relation to early stillbirth.

ELIGIBILITY:
Cases

* Bereaved mothers/parents who have recently birthed a singleton baby who died before/during or immediately after labour between 20 and 28 weeks of pregnancy.
* Baby has no evidence of congenital anomaly
* Able to give written informed consent

Controls

* Pregnant women/people with an ongoing pregnancy (at the target gestation) receiving antenatal care from a participating maternity unit, at a gestation matched to the distribution of stillbirths between 20 to 28 weeks of pregnancy in the same unit
* Baby has no evidence of congenital anomaly
* Able to give written informed consent

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women who have experienced an early stillbirth and women who have an ongoing pregnancy at gestations matched to the profile of women who experienced an early stillbirth from participating maternity units in the UK.
Sampling Method: Probability Sample
Enrollment: 948 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Maternal sleep position during pregnancy | The night prior to questionnaire or the night prior to pregnancy loss
  Self-reported sleep position
Duration of sleep during pregnancy | The night prior to questionnaire or the night prior to pregnancy loss
  Self-reported duration of sleep
Presence of snoring during pregnancy | The night prior to questionnaire or the night prior to pregnancy loss
  Self-reported presence of snoring during pregnancy

SECONDARY OUTCOMES:
Maternal perception of fetal movement frequency | Two-weeks prior to questionnaire or two weeks prior to pregnancy loss
  Self-reported perception of frequency of fetal activity
Maternal perception of fetal movement strength | Two-weeks prior to questionnaire or two weeks prior to pregnancy loss
  Self-reported perception of strength of fetal activity
Maternal caffeine exposure | One month prior to questionnaire
  Self-reported intake of caffeinated drinks
Engagement with antenatal care | Duration of Pregnancy (from booking to the time interview)
  Number of appointments with health professionals
Exposure to Intimate Partner Violence | Duration of Pregnancy (from booking to the time interview)
  Self-reported exposure to abusive behaviour using standardised questions

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Awaiting clearance from the Health Research Authority to share anonymised data for IPD.

REFERENCES:
- [Derived] Heazell AE, Wilkinson J, Morris RK, Simpson N, Smith LK, Stacey T, Storey C, Higgins L. Mothers working to prevent early stillbirth study (MiNESS 20-28): a case-control study protocol. BMJ Open. 2024 Jan 18;14(1):e082835. doi: 10.1136/bmjopen-2023-082835. PMID 38238057

DOCUMENTS (1):
  • Study Protocol (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT06005272/Prot_001.pdf